CLINICAL TRIAL: NCT03060161
Title: Health in the Right Measure: Promoting Healthy Food and Regular Physical Activity Practice for UFRJ Server
Brief Title: Health in the Right Measure: Promoting Healthy Food and Regular Physical Activity Practice for UFRJ Servers
Acronym: HRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Vanessa Chaia Kaippert, Doctor, Universidade Federal do Rio de Janeiro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 123456 CEP
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Human
Keywords: Health promotion; Healthy Diet; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Health

STUDY DESIGN:
Intervention Model Description: The present project corresponds to a longitudinal study. Intervention will be performed soon after the initial diagnosis, through nutritional monitoring and individual guidance on regular physical exercise for a period of 12 weeks. Participants will be evaluated for weight loss, body fat reduction, changes in laboratory parameters and eating habits and in relation to the routine of physical activities immediately after the intervention period, and will be retested after six months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health in the right measure (Experimental): Nutrition counseling and guidance for regular physical activity. An individualized physical exercise program will be proposed according to each participant's level of physical activity and health conditions.
  Participants will also receive individualized nutritional guidance. Throughout the project, collective motivational activities will be carried out to promote healthy eating (culinary workshops, talk wheels and others) and individual activities with all participants, in order to evaluate the adherence of nutritional guidelines and to exchange experiences among them.
  Interventions: Behavioral: Health in the right measure

INTERVENTIONS:
Behavioral: Health in the right measure — Nutritional monitoring and individual guidance on regular physical exercise.

SUMMARY:
Introduction: The epidemiological transition is one of the factors related to the increase in the prevalence of chronic noncommunicable diseases (CNCD), such as cardiovascular diseases, diabetes and cancer. Among the risks of risk to the development of CNCD are obesity, smoking, alcoholism, sedentary lifestyle and inadequate eating habits, with the last two levels having a high impact on gender and disease progression. Objectives: To promote healthy eating habits and to combat physical inactivity through nutritional monitoring and regular physical exercise, using a competition to stimulate adherence of the institution's employees. Methods: The present project is in agreement with the longitudinal study with the work of evaluation (anthropometric, body composition, laboratory and food consumption), in the eats of the times (at the beginning and end of the four-month intervention period). According to nutritional monitoring and individual guidance on regular physical exercise practice over a period of 12 weeks. Weight reduction, body fat reduction, changes in working methods and eating habits, and the relationship to routine physical activity after the intervention period, and are retested after six months. Expected results: Reduction of sedentary lifestyle, weight loss and body fat, improvement of eating habits, quality of life without working environment and health condition of the participants.

DETAILED DESCRIPTION:
The initial goal of the project is to serve approximately thirty UFRJ servers at each edition. The project will be developed in up to two annual editions over a period of five years. After the selection of the candidates, an ambitious meeting will be held with all the participants in order to clarify the objectives and the other stages of the project.

Participants will then be scheduled for laboratory tests and consultations for medical evaluation (exercise test), nutritional assessment and physical evaluation. The anthropometric evaluation will be performed according to previously established protocols. Measurements of body weight, height and waist, abdominal, neck and hip circumference will be performed. The evaluation of the body composition will be performed using the multi-frequency electrical bioimpedance apparatus (Biodynamics® model 450). The usual food consumption quality will be evaluated through dietary records of 3 days (typical 2 days and 1 atypical). In order to evaluate the possible changes in the routine of physical activity practice, the international physical activity questionnaire (IPAQ) will be used in short form. The nutritional consultations will be carried out by nutritionists in the Nutritional Assessment Laboratory (NAL) of the Josué de Castro Nutrition Institute (JCNI).

Blood samples will be collected at the Laboratory of Clinical Analysis of the Faculty of Pharmacy of UFRJ or at the Clinical Pathology Service of the University Hospital Clementino Fraga Filho by properly trained personnel with disposable materials. Blood samples will be collected after a 12 hour fasting for analysis of the complete blood count, lipidogram, liver enzymes (aspartate transaminase and alanine transaminase), glycemia, glycated hemoglobin, free thyroxine and thyroid stimulating hormone.

After performing these evaluations, an individualized physical exercise program will be proposed according to each participant's level of physical activity and health conditions. Participants will also receive individualized nutritional guidance. In case of failure in the stress test the participant will not be able to participate in the physical exercise program, however, he will be invited to remain in activities aimed at promoting healthy eating habits.

Throughout the project, collective motivational activities will be carried out to promote healthy eating (culinary workshops, talk wheels and others) and individual activities with all participants, in order to evaluate the adherence of nutritional guidelines and to exchange experiences among them.

At the end of the project intervention period (12 weeks), the participants will again be submitted to laboratory examination and nutritional assessment: anthropometric and body composition evaluation and evaluation of changes in eating habits.

A collective closure meeting will be held at the end of the project intervention stage and all participants will be informed and will have access to the results of their evaluations to date.

In the next six months participants will be invited to monthly motivational collective activities (sporting challenges, conversation wheel, culinary workshop) as a way to stimulate them to maintain routine physical activities and changes in eating habits.

At the end of three months after the end of the intervention period (6 months of follow-up), the participants will be submitted to nutritional assessment. At the end of the six months after the end of the intervention period, the participants will be submitted to the same evaluations performed three months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Be a server of UFRJ
* Be able to practice some regular physical activity
* Be willing to participate in the proposed activities.

Exclusion Criteria:

* N/A

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Promote healthy eating habits | baseline, after 3 and 9 months
  Changes in dietary habits will be assessed by completing dietary records for three days
Combat physical inactivity | baseline, after 3 and 9 months
  Changes in routine physical activity will be assessed through the International Physical Activity Questionnaire (IPAQ) in the short form.

SECONDARY OUTCOMES:
Effects of lifestyle change on body weight | baseline, after 3, 6 and 9 months
  Changes in body weight will be evaluated.
Effects of lifestyle change on body circumference | baseline, after 3, 6 and 9 months
  Changes in body circumference will be evaluated.
Effects of lifestyle change on body composition | baseline, after 3, 6 and 9 months
  Changes in body composition will be evaluated by electrical bioimpedance
Effects of lifestyle change on biomarkers. | baseline, after 3 and 9 months
  Lipid and glycemic profile will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Eliane Oliveira, Doctor, Principal Investigator — adjunct professor
Locations (1):
- Vanessa Chaia Kaippert, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferreira VA, Magalhaes R. [Nutrition and health promotion: recent perspectives]. Cad Saude Publica. 2007 Jul;23(7):1674-81. doi: 10.1590/s0102-311x2007000700019. Portuguese. PMID 17572817
- [Background] Flegal KM, Shepherd JA, Looker AC, Graubard BI, Borrud LG, Ogden CL, Harris TB, Everhart JE, Schenker N. Comparisons of percentage body fat, body mass index, waist circumference, and waist-stature ratio in adults. Am J Clin Nutr. 2009 Feb;89(2):500-8. doi: 10.3945/ajcn.2008.26847. Epub 2008 Dec 30. PMID 19116329
- [Background] Kyle UG, Bosaeus I, De Lorenzo AD, Deurenberg P, Elia M, Manuel Gomez J, Lilienthal Heitmann B, Kent-Smith L, Melchior JC, Pirlich M, Scharfetter H, M W J Schols A, Pichard C; ESPEN. Bioelectrical impedance analysis-part II: utilization in clinical practice. Clin Nutr. 2004 Dec;23(6):1430-53. doi: 10.1016/j.clnu.2004.09.012. PMID 15556267
- [Background] Lukaski HC, Johnson PE, Bolonchuk WW, Lykken GI. Assessment of fat-free mass using bioelectrical impedance measurements of the human body. Am J Clin Nutr. 1985 Apr;41(4):810-7. doi: 10.1093/ajcn/41.4.810. PMID 3984933
- [Background] Sookoian S, Pirola CJ. Genetics of the cardiometabolic syndrome: new insights and therapeutic implications. Ther Adv Cardiovasc Dis. 2007 Oct;1(1):37-47. doi: 10.1177/1753944707082702. PMID 19124394
- [Background] Obesity: preventing and managing the global epidemic. Report of a WHO consultation. World Health Organ Tech Rep Ser. 2000;894:i-xii, 1-253. PMID 11234459
- [Background] Physical status: the use and interpretation of anthropometry. Report of a WHO Expert Committee. World Health Organ Tech Rep Ser. 1995;854:1-452. PMID 8594834
- [Background] Zeyda M, Stulnig TM. Obesity, inflammation, and insulin resistance--a mini-review. Gerontology. 2009;55(4):379-86. doi: 10.1159/000212758. Epub 2009 Apr 8. PMID 19365105